CLINICAL TRIAL: NCT00632775
Title: Randomized, Double Blind, Controlled Trial of 0.9% NaCl/Dextrose 5% vs 0.45% NaCl/Dextrose 5% as Maintenance Intravenous Fluids in Hospitalized Children
Brief Title: 0.9% NaCl/Dextrose 5% vs 0.45% NaCl/Dextrose 5% as Maintenance Intravenous Fluids in Hospitalized Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Denis Geary, Nephrologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000011114
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Hyponatremia
Keywords: pediatrics; Hyponatremia; Sodium Chloride; maintenance fluids
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subjects in this arm will receive hypotonic (0.45% NaCl/5% dextrose) intravenous (IV) maintenance fluids.
  Interventions: Drug: Hypotonic (0.45% NaCl/5% dextrose) IV maintenance fluids
- 2 (Active Comparator): Subjects in this arm will receive isotonic (0.9% NaCl/5% dextrose) intravenous (IV) maintenance fluids.
  Interventions: Drug: Isotonic (0.9% NaCl/5% dextrose) IV maintenance fluids

INTERVENTIONS:
Drug: Hypotonic (0.45% NaCl/5% dextrose) IV maintenance fluids — Total daily fluid infusion equal to:
  100 mls/kg/day for children weighing <10kg, 1000 mls + 50mls/kg for those weighing 10 to 20 kg, and 1500 mls +20 mls/kg for those >20kg.
  Other Names: 0.45% Sodium Chloride/5% dextrose
  Arms: 1
Drug: Isotonic (0.9% NaCl/5% dextrose) IV maintenance fluids — Total daily fluid infusion equal to:
  100 mls/kg/day for children weighing <10kg, 1000 mls + 50mls/kg for those weighing 10 to 20 kg, and 1500 mls +20 mls/kg for those >20kg.
  Other Names: 0.9% Sodium Chloride/5% Dextrose
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the mean serum sodium at 48 hours following the initiation of therapy with either 0.45% NaCl/dextrose 5% or 0.9% NaCl/dextrose 5%, in children requiring maintenance IV fluid administration.

DETAILED DESCRIPTION:
Hyponatremia, has become increasingly recognized as a cause of morbidity and mortality in hospitalized children. The main etiology of hyponatremia in these children has been attributed to the use of hypotonic maintenance IV fluids. The practice of providing IV solutions containing 20-30 mmol/L of Na is based on "physiological needs" proposed by Holliday and Segarin 1957, derived from studies of 61 adults and children. The presence of non-physiologic ADH secretion in the great majority of hospitalized children due to nausea, stress, pain, and surgical interventions, has confirmed that Holliday and Segar's recommendations are frequently inappropriately applied. To avoid the development of hyponatremia, it has been suggested that isotonic 0.9% NaCl/dextrose 5% should be the standard maintenance IV solution.

The routine use of an isotonic maintenance fluid solution has not yet been studied, and concerns exist regarding the potential for hypernatremia and salt and water overload. If isotonic solutions are to be recommended routinely, their overall safety, and specifically the occurrence of dysnatremias and volume overload, should be evaluated in a controlled prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 month to 18 years
* Anticipated hospitalization >48 hours
* Initial plasma Na between 135-145 mmol/L, with a management plan(determined by the responsible physician) to include IV fluids at > 80% of maintenance
* For children who have had an IV saline bolus, it must have been completed three or more hours prior to having baseline bloods
* Baseline bloods must be drawn within 3 hours of initial patient contact.

Exclusion Criteria:

* Diagnosed with, or clinically suspected to have, any of the following: dehydration/gastroenteritis, heart or liver failure, portal hypertension with ascites, metabolic disease, SIADH, diabetes insipidus or mellitus, hypertension, adrenal insufficiency, renal failure [creatinine>100 μmol/L (<3 years); >150 μmol/L (> 3 years)], nephritic or nephrotic syndrome, Kawasaki disease, Sickle cell disease if requiring hyperhydration.
* Clinically edematous
* On diuretic medications
* Plasma glucose is >15 mmol/L
* Require CCU admission
* Any patients requiring IV maintenance therapy having conditions/diseases not listed as excluded are eligible to be in this study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2007-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma urea, creatinine, glucose and electrolyte levels | At the time of IV start and every 24 hours thereafter

SECONDARY OUTCOMES:
Oral fluid intake | The duration of the patient's participation in the study
Weight | Every 24 hours
Standardized clinical assessment of edema | Every 24 hours
Blood pressure | Every morning

CONTACTS AND LOCATIONS:
Overall Officials: Denis Geary, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Friedman JN, Beck CE, DeGroot J, Geary DF, Sklansky DJ, Freedman SB. Comparison of isotonic and hypotonic intravenous maintenance fluids: a randomized clinical trial. JAMA Pediatr. 2015 May;169(5):445-51. doi: 10.1001/jamapediatrics.2014.3809. PMID 25751673